CLINICAL TRIAL: NCT04527861
Title: Oncologic Outcomes of Single-incision Laparoscopic Surgery Versus Conventional Laparoscopic Surgery for Colorectal Cancer: A Multi-center, Prospective, Open Label, Non-inferiority, Randomized Controlled Trial
Brief Title: Oncologic Outcomes of Single-incision Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Acronym: CSILS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Dongfang Hospital Affiliated to Tongji University (Other); Fudan University (Other); Changhai Hospital (Other); Shengjing Hospital (Other); RenJi Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Zhejiang Provincial People's Hospital (Other); Shandong Provincial Hospital (Other Government); The General Hospital of Western Theater Command (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhao Ren, Chief Physicion, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSILS
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectal Cancer
Keywords: single-incision laparoscopic surgery; conventional laparoscopic surgery; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-incision Laparoscopic Surgery (Experimental): Patients with colorectal cancer undergo single-incision laparoscopic surgery.
  Interventions: Procedure: Single-incision Laparoscopic Surgery
- Conventional Laparoscopic Surgery (Active Comparator): Patients with colorectal cancer undergo conventional laparoscopic surgery（3~5 ports）.
  Interventions: Procedure: Conventional Laparoscopic Surgery

INTERVENTIONS:
Procedure: Single-incision Laparoscopic Surgery — In this group，the surgery is performed through a single incision. The surgeon will adjust surgical position to expose the operative field with the help of gravity. Besides，hand over hand cross and parallel techniques are needed to achieve the SILS. All the other operative procedures are the same as conventional laparoscopic surgery.
  Other Names: SILS
  Arms: Single-incision Laparoscopic Surgery
Procedure: Conventional Laparoscopic Surgery — In this group，the surgery is performed through 3-5 ports according to the surgeons habits and specific conditions.
  Other Names: CLS
  Arms: Conventional Laparoscopic Surgery

SUMMARY:
This study is designed to investigate long-term oncologic outcomes of single-incision laparoscopic surgery (SILS) compared to conventional laparoscopic surgery (CLS) for colorectal cancer.

DETAILED DESCRIPTION:
In order to improve cosmetic effect and reduce postoperative pain, single-incision laparoscopic surgery (SILS) is attracting increasing attention. SILS is considered to be the next major advance in the progress of minimally invasive surgical approaches to colorectal disease that is more feasible in generalized use. In most previous studies, SILS for colorectal cancer was feasible and short-term safe compared to conventional laparoscopic surgery (CLS) . However, there is still controversy over its potential better cosmetic effect and less postoperative pain. Moreover, the long-term oncologic outcomes are still inconclusive as only a few studies showed long-term survival data. Up to now, most studies were limited to their retrospective nature and small samples. So more studies, especially large-scale, randomized controlled trials are needed to establish the best indications for SILS for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age ≤85 years
* Tumor located in colon and high rectum ( the lower border of the tumor is above the peritoneal reflection)
* Pathological or highly suspected colorectal carcinoma
* Clinically diagnosed cT1-4aN0-2 M0 lesions according to the 8th Edition of AJCC Cancer Staging Manual
* Tumor size of 5 cm or less
* ECOG score is 0-1
* ASA score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Body mass index (BMI) >35 kg/m2
* The lower border of the tumor is located distal to the peritoneal reflection
* Familial adenomatous polyposis (FAP)
* Inflammatory bowel disease (IBD)
* Multiple malignant colorectal tumors
* Pregnant woman or lactating woman
* Severe mental disease
* Previous gastrointestinal surgery (except appendectomy ）
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by colorectal cancer
* Requirement of simultaneous surgery for other disease
* Simultaneous or metachronous multiple cancers with disease-free survival ≤ 5 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months after surgery
  3-year disease free survival rate

SECONDARY OUTCOMES:
Operative time | intraoperative
  Operative time（minutes）
Intraoperative blood loss | intraoperative
  Estimated blood loss（milliliters，ml）
Incision length | intraoperative
  Incision length（centimeters，cm）
Total incision length | intraoperative
  The sum of all incision lengths（centimeters，cm）
Conversion rate | intraoperative
  The proportion of converted to laparotomy and added trocars（%）
Length of stay | 1-14 days after surgery
  The postoperative day when patients complied with the predefined discharge criteria（days after surgery）
Postoperative recovery course | 1-14 days after surgery
  Time to first ambulation, flatus, liquid diet and semi-liquid diet （hours after surgery）
Early morbidity rate | 30 days after surgery
  morbidity rate 30 days after surgery
Pain score | 1-3 days after surgery
  Postoperative pain is recorded using the visual analog scale (VAS) pain score （0-10 points）tool on postoperative day 1, 2, 3
Tumor size | 14 days after surgery
  The diameter of tumors（centimeters，cm）
Incisal margin | 14 days after surgery
  Length of proximal and distal margin （centimeters，cm）
Lymph node detection | 14 days after surgery
  Lymph nodes harvested（numbers）
Cosmetic effect | 1 month, 6 months and 1 year after surgery
  Assessed using a "Beauty Questionnaire" evaluating patient's satisfaction according to a 5-scale score, ranging from ''Not satisfied at all'' to ''Very satisfied''
The quality of life-Core | 1 month, 6 months and 1 year after surgery
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
The quality of life-Colorectal | 1 month, 6 months and 1 year after surgery
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal 29 (EORTC QLQ-CR29)
5-year overall survival rate | 60 months after surgery
  5-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, MD, PHD, Principal Investigator — Ruijin Hospitlal , Shanghai Jiaotong University School of Medicine; Chun Song, MD, Study Director — Dongfang Hospital Affiliated to Tongji University; Ye Xu, MD, Study Director — Shanghai Cancer Center; Liqiang Hao, MD, Study Director — Changhai Hospital; Hong Zhang, MD, Study Director — Shengjing Hospital; Hong Zhou, MD, Study Director — RenJi Hospital; Qingtong Zhang, MD, Study Director — Liaoning Cancer Hospital & Institute; Shiliang Tu, MD, Study Director — Zhejiang Provincial People's Hospital; Xiaoqiao Zhang, MD, Study Director — Shandong Provincial Hospital; Lin Zhang, MD, Study Director — The General Hospital of Western Theater Command; Feng Gao, MD, Study Director — The 940th Hospital of Joint Logistic Support Force of Chinese of PLA
Locations (11):
- China (11):
  - The 940th Hospital of Joint Logistic Support Force of Chinese of PLA, Lanzhou, Gansu
  - Shengjing Hospital, Shenyang, Liaoning
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The General Hospital of Western Theater Command, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Shanghai Cancer Center, Shanghai
  - Dongfang Hospital Affiliated to Tongji University, Shanghai
  - RenJi Hospital, Shanghai
  - Changhai Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maggiori L, Tuech JJ, Cotte E, Lelong B, Denost Q, Karoui M, Vicaut E, Panis Y. Single-incision Laparoscopy Versus Multiport Laparoscopy for Colonic Surgery: A Multicenter, Double-blinded, Randomized Controlled Trial. Ann Surg. 2018 Nov;268(5):740-746. doi: 10.1097/SLA.0000000000002836. PMID 30303873
- [Background] Lee YS, Kim JH, Kim HJ, Lee SC, Kang BM, Kim CW, Lim SW, Lee SH, Kim JG. Short-term Outcomes of Single-port Versus Multiport Laparoscopic Surgery for Colon Cancer: The SIMPLE Multicenter Randomized Clinical Trial. Ann Surg. 2021 Feb 1;273(2):217-223. doi: 10.1097/SLA.0000000000003882. PMID 32209897
- [Derived] Song Z, Liu K, Zhang T, Wang B, Shi Y, Jiang Y, Wang C, Chen X, Ji X, Zhao R. Oncologic outcomes of single-incision laparoscopic surgery versus conventional laparoscopic surgery for colorectal cancer (CSILS): study protocol for a multicentre, prospective, open-label, noninferiority, randomized controlled trial. BMC Cancer. 2022 Jul 7;22(1):743. doi: 10.1186/s12885-022-09821-9. PMID 35799145